CLINICAL TRIAL: NCT00616408
Title: Predictive Value of 3 Months Results on 12 Months Tumor Shrinkage After First-Line Octreotide-LAR Therapy in Patients With Acromegaly
Brief Title: Prediction of Tumor Shrinkage in Acromegaly
Status: Completed | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Annamaria Colao, Department of Molecular and Clinical Endocrinology and Oncology University Federico II of Naples
Other Study IDs: NeuroendoUnit-8
Record Dates: First submitted 2008-02-05; First posted 2008-02-15 (Estimated); Last update posted 2008-02-15 (Estimated); Status verified 2007-12

CONDITIONS: Acromegaly
Keywords: GH; IGF-I; GH-secreting tumors; Octreotide
MeSH Terms: conditions — Acromegaly | interventions — Octreotide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A: Newly diagnosed active acromegaly out of the 297 patients coming to our Department for acromegaly who received first-line treatment with LAR
  Interventions: Drug: Octreotide-LAR

INTERVENTIONS:
Drug: Octreotide-LAR — Initial dose is 20 mg every 28 d for three months, then the dose is down-titrated to 10 mg/q28d if GH levels are below 1 ng/ml, up-titrated to 30 mg/q28d if GH levels are above 10 ng/ml and remains to 20 mg/q28 d if GH is between 1-10 ng/ml
  Other Names: Sandostatin (Novartis Pharma)

SUMMARY:
In the last two decades, somatostatin analogs have become a cornerstone of medical therapy for acromegaly. One year of treatment with octreotide-LAR (LAR) controls GH and IGF-I excess in 54% and 63% of unselected patients, with an increasing proportion of subjects achieving IGF-I normalization prolonging the treatment. Clinically significant tumor shrinkage (20-30% vs. baseline) has also been reported, with a higher proportion in patients treated first-line [231 of 448 patients (52%)] than in those treated after surgery and/or radiotherapy [52 of 248 patients (21%)]. The highest rate of clinically significant shrinkage (>20%) occurred in patients treated first-line with LAR (80%) as compared to the short-lasting octreotide formulation (50%) or lanreotide slow-release formulation (35%. In 99 de novo patients with acromegaly, we recently reported control of GH levels in 57.6%, of IGF-I levels in 45.5% and a greater than 50% tumor shrinkage in 44.4% after 12 months of first-line treatment with somatostatin analogues, either LAR or lanreotide. Besides the different drug used, the duration of treatment also plays an important role on the shrinkage magnitude. In a homogeneous cohort of 56 patients treated with LAR only and continuously for 24 months, we noted an even more sustained effect on tumor shrinkage: overall, tumor volume decreased by 68.1±16.5% using dosages up-titrated to 40 mg every 28 days.

Despite this evidence, there is still a debate on the use of first-line treatment with somatostatin analogues. Of paramount importance would be the possibility to predict the results of one year treatment early after treatment beginning. Controversy has been reported on the predictive value of initial tumor size, inhibition of GH and IGF-I levels during treatment, and dose or type of the somatostatin analogue used during treatment. We found that percent suppression of IGF-I after 12 months of LAR treatment was the parameter that best predicted the amount of tumor shrinkage after the same period, but did not investigate the results of short-term treatment in the same series.

This observational, analytical, open, retrospective study was designed to evaluate the predictive value of tumor shrinkage, GH and IGF-I suppression after 3 months of Octreotide-LAR (LAR) on tumor shrinkage obtained after 12 months. As secondary parameters we also studied baseline patients profile such as age of diagnosis, gender, estimated disease duration, GH and IGF-I levels and tumor size.

DETAILED DESCRIPTION:
From Jan 1st 1995 to December 31st 2006, all files of patients with newly diagnosed active acromegaly out of the 297 patients coming to our Department for acromegaly who received first-line treatment with LAR will be considered for this study.

As our routine procedure, all patients signed an informed consent to approve diagnostic testing, treatment decision, methods for follow-up and data treatment for scientific purposes. This study has been conducted in accordance with the Helsinki II Declaration on human experimentation. This study takes advantage from data collected in a large, prospective study to investigate the effect of first-line surgery or medical therapy (with somatostatin analogues and/or dopamine/agonists) on GH, IGF-I, tumor mass, cardiovascular risk markers, cardiomyopathy, hypertension, metabolic profile and prostate diseases in all the patients coming for a diagnosis of acromegaly in our Department and approved by our Ethical Committee the 14/10/97 (no.60/97).

ELIGIBILITY:
Inclusion Criteria:

* No previous treatment for acromegaly

Exclusion Criteria:

* primary surgery
* concomitant hyperprolactinemia requiring combined somatostatin analogues and dopamine-agonist treatment
* primary treatment with lanreotide

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed patients with acromegaly treated first-line with octreotide-LAR
Sampling Method: Probability Sample
Enrollment: 61 (Actual)
Dates: Start 1997-01; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
GH and IGF-I age-normalized levels, percent GH and IGF-I suppression and percent tumor shrinkage after 3 months | 12 months

SECONDARY OUTCOMES:
baseline age, gender, estimated disease duration, GH and IGF-I levels, tumor size | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Annamaria Colao, MD, Principal Investigator — University Federico II of Naples
Locations (1):
- Department of Molecular and Clinical Endocrinology and Oncology, University Federico II of Naples, Naples, Italy

REFERENCES:
- [Result] Colao A, Pivonello R, Auriemma RS, Galdiero M, Savastano S, Lombardi G. Beneficial effect of dose escalation of octreotide-LAR as first-line therapy in patients with acromegaly. Eur J Endocrinol. 2007 Nov;157(5):579-87. doi: 10.1530/EJE-07-0383. PMID 17984237
- [Result] Mercado M, Borges F, Bouterfa H, Chang TC, Chervin A, Farrall AJ, Patocs A, Petersenn S, Podoba J, Safari M, Wardlaw J; SMS995B2401 Study Group. A prospective, multicentre study to investigate the efficacy, safety and tolerability of octreotide LAR (long-acting repeatable octreotide) in the primary therapy of patients with acromegaly. Clin Endocrinol (Oxf). 2007 Jun;66(6):859-68. doi: 10.1111/j.1365-2265.2007.02825.x. Epub 2007 Apr 25. PMID 17465997
- [Result] Resmini E, Dadati P, Ravetti JL, Zona G, Spaziante R, Saveanu A, Jaquet P, Culler MD, Bianchi F, Rebora A, Minuto F, Ferone D. Rapid pituitary tumor shrinkage with dissociation between antiproliferative and antisecretory effects of a long-acting octreotide in an acromegalic patient. J Clin Endocrinol Metab. 2007 May;92(5):1592-9. doi: 10.1210/jc.2006-2084. Epub 2007 Feb 20. PMID 17311860
- [Result] Colao A, Pivonello R, Auriemma RS, Briganti F, Galdiero M, Tortora F, Caranci F, Cirillo S, Lombardi G. Predictors of tumor shrinkage after primary therapy with somatostatin analogs in acromegaly: a prospective study in 99 patients. J Clin Endocrinol Metab. 2006 Jun;91(6):2112-8. doi: 10.1210/jc.2005-2110. Epub 2006 Mar 14. PMID 16537687
- [Result] Cozzi R, Montini M, Attanasio R, Albizzi M, Lasio G, Lodrini S, Doneda P, Cortesi L, Pagani G. Primary treatment of acromegaly with octreotide LAR: a long-term (up to nine years) prospective study of its efficacy in the control of disease activity and tumor shrinkage. J Clin Endocrinol Metab. 2006 Apr;91(4):1397-403. doi: 10.1210/jc.2005-2347. Epub 2006 Jan 31. PMID 16449332
- [Result] Sheppard MC. Primary medical therapy for acromegaly. Clin Endocrinol (Oxf). 2003 Apr;58(4):387-99. doi: 10.1046/j.1365-2265.2003.01734.x. PMID 12641619
- [Derived] Colao A, Pivonello R, Auriemma RS, Galdiero M, Savastano S, Grasso LF, Lombardi G. Growth hormone-secreting tumor shrinkage after 3 months of octreotide-long-acting release therapy predicts the response at 12 months. J Clin Endocrinol Metab. 2008 Sep;93(9):3436-42. doi: 10.1210/jc.2008-0424. Epub 2008 Jul 1. PMID 18593770